CLINICAL TRIAL: NCT03554772
Title: A Randomized, Double-Blind, Placebo-Controlled, Efficacy, Tolerability, Safety and Pharmacokinetic Study of Single Doses of DFN-15 in Post-Surgical Dental Pain
Brief Title: Efficacy, Tolerability, Safety, and Pharmacokinetic Study of DFN-15
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFN-15-CD-010
Record Dates: First submitted 2018-05-21; First posted 2018-06-13 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-08

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DFN-15 (Celecoxib Oral Solution) 62.5 mg (Experimental): Single dose containing 62.5 mg of celecoxib in 10 ml solution
  Interventions: Drug: DFN-15 (Celecoxib Oral Solution) 62.5 mg
- DFN-15 (Celecoxib Oral Solution) 125 mg (Experimental): Single dose containing 125 mg of celecoxib in 10 ml solution
  Interventions: Drug: DFN-15 (Celecoxib Oral Solution) 125 mg
- DFN-15 (Celecoxib Oral Solution) 250 mg (Experimental): Single dose containing 250 mg of celecoxib in 10 ml solution
  Interventions: Drug: DFN-15 (Celecoxib Oral Solution) 250 mg
- Placebo (Placebo Comparator): Single dose containing 0 mg of celecoxib in 10 ml solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DFN-15 (Celecoxib Oral Solution) 62.5 mg — Oral Solution
  Arms: DFN-15 (Celecoxib Oral Solution) 62.5 mg
Drug: DFN-15 (Celecoxib Oral Solution) 125 mg — Oral Solution
  Arms: DFN-15 (Celecoxib Oral Solution) 125 mg
Drug: DFN-15 (Celecoxib Oral Solution) 250 mg — Oral Solution
  Arms: DFN-15 (Celecoxib Oral Solution) 250 mg
Drug: Placebo — Oral Solution
  Arms: Placebo

SUMMARY:
Efficacy, Tolerability, Safety and Pharmacokinetic Study of DFN-15 in Post-Surgical Dental Pain.

DETAILED DESCRIPTION:
This is a Phase 2, single-center, randomized, double blind, dose-ranging placebo-controlled, clinical study evaluating the efficacy, tolerability, safety, and the pharmacokinetic properties of a known drug (selective COX-2 inhibitor) administered as an alternative formulation/dosage form (DFN-15, a liquid oral formulation) in an accepted model of acute post-operative pain (acute pain following oral surgery for extraction of bilateral impacted mandibular third molar teeth in otherwise healthy subjects).120 female and male healthy subjects scheduled to undergo elective bilateral third molar extraction will be randomized, after they provide informed consent and are confirmed to meet all the study selection criteria, in a 1:1:1:1 ratio to receive a single oral dose of either DFN-15 Dose A DFN-15 Dose B, DFN-15 Dose C or matching placebo.

Subjects will undergo a screening procedure (within 28 days of the scheduled extraction of the impacted third molars) that will involve the collection of demographic information, height, weight and body mass index (BMI), urine pregnancy test (women of child-bearing potential,) medical and medicinal history, physical examination, dental examination, vital signs measurement (blood pressure, pulse rate, respiratory rate), clinical laboratory investigation (hematology,serology, coagulation parameters, serum chemistry and urinalysis),12-lead ECG and a panoramic x-ray to document the impacted mandibular third molar teeth. As a pre-requisite for randomization, subjects will be required to report "moderate" to "severe" baseline pain on the provided paper diary within 6 hours post-surgery (called the 'Baseline' period) as characterized on a 4-point categorical pain intensity (PI) scale (0= none, 1= mild, 2= moderate, 3= severe), and a score of ≥5, on the 11-point Numerical Pain Rating Scale (NPRS) where 0 represents 'no pain' and 10 represents 'worst pain imaginable'. Eligible subjects will be randomized and will receive a single dose of the assigned study treatment. Subjects will be randomized and administered the study medication within 15 minutes of meeting the post-operative inclusion criteria (baseline score).Subjects will be assessed at pre-specified time-points over an observation period of 8 hours from the time of randomization.

Subjects with inadequately controlled pain symptoms may request rescue analgesic medication. Subjects will be encouraged to delay using the rescue medication if their pain is tolerable until 120 minutes post-dose of study medication. A subject who is administered rescue pain medication will continue completing pain assessments until 8 hours after treatment initiation. All randomized subjects will be provided with a paper diary to record pain assessments (Pain Intensity on 11-point NPRS scale, followed by Pain Relief using a 5-point categorical scale [where 0= no pain relief, 1= little pain relief, 2= some pain relief, 3= a lot of pain relief, 4= complete pain relief]) At study medication administration, two stopwatches will be started, to measure times to 'perceptible' and 'meaningful' pain-relief. Subjects will be instructed to stop the first stopwatch when they first perceive pain relief to occur (time to perceptible relief). Subjects will be instructed to stop the second stopwatch when they first experience meaningful pain relief (time to meaningful relief). Stopwatch times of perceptible relief and meaningful relief will be recorded using exact stopwatch time displayed.

In addition, at 8 hours post-dose or within 5 minutes prior to first use of rescue medication (whichever is earlier), subjects will be asked to record within the provided patient diary: 'Patient Rating of Treatment Satisfactoriness' using a 5-point verbal rating scale (0 =poor, 1 =fair, 2 =good, 3=very good, 4 =excellent).

Subjects will remain NPO (nothing by mouth), including water, from Check-in (i.e., at least 2 hours before the administration of the dose of study medication to randomized subjects) until 2 hours post-dose, on Day 1 (study day). After 2 hours post-dose, subjects may be permitted to consume water, or gelatin snacks. Subjects are prohibited from ingesting solid foods or carbonated beverages for at least 6 hours post-dose.

12-lead ECG and Vital Signs were performed before surgery, at baseline and at periodic intervals post-dose until 8 hours .At discharge (8 hours post-randomization) from the clinical facility, all AEs reported for the subjects will be reviewed. A physical examination, including evaluation of the incision site for hematomas, and clinical laboratory evaluation (coagulation parameters and specific hematology, serum biochemistry and urinalysis parameters) will be conducted.

All subjects will have blood drawn at specified time points (pre-dose and over the 8 hour observation period) for pharmacokinetic evaluation.

Subjects will return to the research center 7 days (± 3 days) post-surgery for evaluation of their safety and well-being. Any AEs experienced post-surgery will be reviewed. A physical examination, of the subject will be performed, 12-lead ECG, and vital signs parameters will be repeated. Hematology, coagulation parameters, serum biochemistry and urinalysis parameters will be repeated only if there is a clinically significant abnormality or ongoing AE(s). Any changes to the prior and concomitant medication made after discharge will be reviewed and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled to undergo elective bilateral lower (mandibular) third molar extraction under local anesthesia.
2. Subjects must be generally healthy, ambulatory, able to understand and willing to comply with study procedures, study restrictions, assessments, and requirements per the discretion of the investigator.
3. Subjects must voluntarily sign written informed consent prior to any study-specific procedures.
4. Subjects must have a body mass index (BMI) greater than or equal to 19.0 to less than or equal to 35.0

Exclusion Criteria:

1. History of migraine or frequent headaches, low back pain, or other acute or chronic pain conditions.
2. Acute illness or unresolved local infection prior to surgery that can interfere with the conduct of the study.
3. Positive results on urine drug screen or alcohol breath test indicative of illicit drug (Cocaine Metabolites, Marijuana (THC), MDMA (Ecstasy) and Phencyclidine) or alcohol abuse at screening and/or prior to extraction procedure.
4. Positive results for the following (prescription included): Amphetamines, Barbiturates, Benzodiazepines, Methadone, Methamphetamine, Opiates, Oxycodone, and Tricyclic Antidepressants.
5. Frequent use of nicotine-containing products.
6. Excessive intake of caffeine-containing foods or beverages within 48 hours prior to surgery.
7. Routinely uses pain medication.
8. Currently taking any corticosteroid chronically (except for an inhaled steroid for pulmonary disease, and local topical or ophthalmic steroid) or has taken systemic corticosteroids within 4 weeks of the proposed date of surgery.
9. Currently taking central nervous system active drugs such as hypnotics, sedatives, monoamine oxidase inhibitors, sympathomimetic amines, benzodiazepines, tricyclic antidepressants, or serotonin norepinephrine reuptake inhibitors, and anticonvulsants for pain.
10. Donated blood products or had blood loss greater than 500 mL 30 days prior to Screening or between Screening and surgery.
11. Member or relative of study staff or the Sponsor directly involved in the study.
12. Previous participation in this study.
13. Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 30 days prior to the Screening visit.
14. Currently receiving or have received within 7 days prior to investigational product administration in the study, any drug (s) that is metabolized by hepatic microsomal enzyme CYP 2D6.
15. Clinically significant disease or disorder which may put the subject at risk, influence the results or the subject's ability to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elimor Brand-Schieber, PhD, Study Director — Director-Clinical Development
Locations (1):
- Site 101, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singla N, Bertoch T, Shenoy S, Munjal S. Efficacy and safety of single-dose DFN-15 for treatment of acute postsurgical dental pain: a randomized, double-blind, placebo-controlled study. Pain. 2022 Jan 1;163(1):91-99. doi: 10.1097/j.pain.0000000000002312. PMID 34252915

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | DFN-15 (Celecoxib Oral Solution) 62.5 mg | DFN-15 (Celecoxib Oral Solution) 125 mg | DFN-15 (Celecoxib Oral Solution) 250 mg
Started | 30 | 30 | 29 | 31
Completed Treatment Period (8 Hours Post Dose) | 30 | 30 | 29 | 31
Completed | 30 | 30 | 29 | 29
Not Completed | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DFN-15 (Celecoxib Oral Solution) 62.5 mg | DFN-15 (Celecoxib Oral Solution) 125 mg | DFN-15 (Celecoxib Oral Solution) 250 mg | Total
Number analyzed (Participants) | 30 | 30 | 29 | 31 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (2.70) | 19.6 (2.45) | 19.2 (1.64) | 20.5 (2.45) | 19.8 (2.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 17 | 13 | 60
  Male | 14 | 16 | 12 | 18 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 4 | 7 | 23
  Not Hispanic or Latino | 24 | 24 | 25 | 24 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 0 | 3
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 28 | 26 | 22 | 28 | 104
  More than one race | 0 | 1 | 2 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 2 | 2 | 5
BMI [Mean (Standard Deviation); unit: kg/ m^2] — Body Mass Index is calculated as Weight (in kg)/ Height (in m) ^ 2
  kg/ m^2 | 26.4 (4.15) | 27.1 (5.03) | 25.1 (4.11) | 24.4 (4.41) | 25.8 (4.51)
Qualifying Baseline Categorical Pain Score [Count of Participants; unit: Participants]
  0 = No Pain | 0 | 0 | 0 | 0 | 0
  1= Mild Pain | 0 | 0 | 0 | 0 | 0
  2= Moderate Pain | 8 | 13 | 11 | 12 | 44
  3= Severe Pain | 22 | 17 | 18 | 19 | 76

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Difference Over the First Six Hours
Description: The primary endpoint is the Summed Pain Intensity Difference over the first 6 hours (SPID6) after dosing compared between DFN-15 and placebo. Pain intensity (P) will be measured at timepoints of 15, 30, and 45 minutes and 1, 1.5, 2, 3, 4, 5 and 6, hours after baseline ,using 11-point Pain Intensity Numerical Rating Scale (NPRS). Zero (0) equals no pain and Ten (10) equals worst pain imaginable.
  SPID6 is created by summing the time weighted pain intensity differences (PID) scores using the area under the PID curve methodology. All SPID calculations will be performed using the standard trapezoidal rule SPIDx =∑_(i=0)^x▒((〖PID〗_i+〖PID〗_(i+1))/2) * (T_(i+1)- T_i ) Where: PID_i = P_i - PBL (Pain score at time i and Pain score at Baseline), and (T_i+1 - T_i) is the Time difference in minutes between time i and time i+1.
  Therefore, SPID6 values may theoretically range between a maximum score of 0 ( no improvement) and a minimum score of -3525 (best improvement)
Time Frame: 6 hours post dose
Population: mITT Population : defined as all randomized subjects who received study drug and recorded at least one post-dosing PI score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | DFN-15 (Celecoxib Oral Solution) 62.5 mg | DFN-15 (Celecoxib Oral Solution) 125 mg | DFN-15 (Celecoxib Oral Solution) 250 mg
Number analyzed (Participants) | 30 | 30 | 29 | 31
units on a scale | -420.2 (716.42) | -1101.0 (570.74) | -1771.7 (646.10) | -1463.5 (727.28)
Statistical Analysis 1: Comparison: Placebo vs DFN-15 (Celecoxib Oral Solution) 62.5 mg vs DFN-15 (Celecoxib Oral Solution) 125 mg vs DFN-15 (Celecoxib Oral Solution) 250 mg; Test type: Superiority; p < 0.0001, ANCOVA — p-value for each dose group vs placebo comparison; ANCOVA model included treatment as main effect , baseline NPRS and basline BMI as covariates P-value is Dunnett adjusted (individual treatment arms)

ADVERSE EVENTS:
Time Frame: All AEs, whether volunteered, elicited, or noted on physical examination, and regardless of causality or seriousness, were assessed and recorded in the CRF beginning after administration of study drug through the final follow-up assessment (approximately 7 ± 3 days after the last study drug administration). Additionally, if the investigator became aware of the occurrence of an SAE within 30 days of the last visit, the SAE was reported.
Arm/Group | Placebo | DFN-15 (Celecoxib Oral Solution) 62.5 mg | DFN-15 (Celecoxib Oral Solution) 125 mg | DFN-15 (Celecoxib Oral Solution) 250 mg
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 4/30 | 5/30 | 4/29 | 5/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | DFN-15 (Celecoxib Oral Solution) 62.5 mg (N=30) | DFN-15 (Celecoxib Oral Solution) 125 mg (N=29) | DFN-15 (Celecoxib Oral Solution) 250 mg (N=31)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Urine Present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerular Filtration Rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International Normalized Ratio increaed (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alveolar Osteitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT03554772/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03554772/SAP_001.pdf